CLINICAL TRIAL: NCT03680326
Title: Influence of Intravitreal Anti-vascular Endothelial Growth Factor Administration on Vitreomacular Interface- and Retinal Morphology in Eyes With Neovascular Age-related Macular Degeneration
Brief Title: Intravitreal Anti-vascular Endothelial Growth Factor Administration and Its Influence on Vitreomacular Interface- and Retinal Morphology in Eyes With Neovascular Age-related Macular Degeneration
Status: Completed | Type: Observational
Sponsor: Hospital Hietzing (Other)
Responsible Party: Principal Investigator, Dr. Clara Wernigg, Dr., Hospital Hietzing
Other Study IDs: Interface, vitreomacular
Record Dates: First submitted 2018-09-17; First posted 2018-09-21 (Actual); Last update posted 2018-09-21 (Actual); Status verified 2018-09

CONDITIONS: Vitreomacular Interface

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- OCT: only optical coherence tomography and visual acuity testing at each visit, patients were recruited retrospectively, only data analysis
  Interventions: Device: OCT

INTERVENTIONS:
Device: OCT — only OCT

SUMMARY:
Purpose:

To assess the influence of intravitreal anti-vascular endothelial growth factor (anti-VEGF) administration on vitreomacular interface- and retinal morphology in eyes with neovascular age-related macular degeneration (AMD) and to identify morphological markers potentially influencing disease prognosis.

Methods:

43 patients (51 eyes) with treatment naïve neovascular AMD subsequently treated with Bevacizumab 1.25mg (in 0.05ml of solution) were monitored until month 12 of follow-up. Following a loading dose of 3 monthly intravitreal anti-VEGF injections, patients were treated as-needed [pro re nata (PRN)]. Functional and morphological changes were assessed using Spectral Domain Optical Coherence Tomography (SD-OCT).

DETAILED DESCRIPTION:
This retrospective study included 43 treatment-naive patients (51 eyes) with neovascular AMD over the course of 12 months. Patients were treated with a loading dose of 3 initial monthly anti-VEGF injections (Bevacizumab 1.25mg in 0.05ml of solution-Avastin®) and were followed monthly until year 1. Re-treatment was performed if needed (pro re nata-PRN) as previously reported.

ELIGIBILITY:
Inclusion Criteria:

- diagnosis of treatment-naive neovascular AMD

Exclusion Criteria:

* any treatment with other anti-VEGF agents than Bevacizumab in the follow-up period
* any other diseases leading to macular edema
* prior vitrectomy
* uveitis
* retinal or corneal laser surgery
* high myopia (>6dpt)
* preceding eye trauma

Ages: 66 Years to 98 Years | Sex: All
Age Groups: Older Adult
Study Population: treatment-naive patients with neovascular AMD
Sampling Method: Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2015-02-02 (Actual); Primary Completion 2018-03-22 (Actual); Study Completion 2018-04-14 (Actual)

PRIMARY OUTCOMES:
visual acuity | 12 months
  visual acuity testing was performed

IPD SHARING:
Plan to Share IPD: No